CLINICAL TRIAL: NCT04247243
Title: Streamlining Care Delivery in the Paediatric Emergency Department Using Rapid Point-of-care Diagnostics for Group a Streptococcus: a Randomized Controlled Trial
Brief Title: Rapid POC GAS Diagnostics in the Paediatric ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HAHSO POC GAS
Record Dates: First submitted 2020-01-20; First posted 2020-01-30 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-03

CONDITIONS: Streptococcal Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Rapid testing (Experimental): Abbott ID NOW Strep A testing.
  Interventions: Device: Rapid testing
- Reference testing (Active Comparator): Culture-based testing.
  Interventions: Diagnostic Test: Reference testing

INTERVENTIONS:
Device: Rapid testing — Abbott ID NOW Strep A testing
  Arms: Rapid testing
Diagnostic Test: Reference testing — Culture-based testing
  Arms: Reference testing

SUMMARY:
Randomized trial evaluating effectiveness of rapid point-of-care molecular GAS diagnostics as compared to standard culture-based techniques for the management of children aged 3-18 years of age presenting with sore throat to McMaster Children's Hospital Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* all those presenting who have a throat swab ordered for GAS testing

Exclusion Criteria:

* those who took antibiotics effective against GAS within 72 h of ED presentation

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 392 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Appropriate antibiotic treatment | 3-5 days post-enrolment
  All participants will be contacted by phone to ascertain whether they took antibiotics for the treatment of streptococcal pharyngitis. 'Appropriate antibiotic treatment' is a dichotomous measure. If the participant's throat swab was positive for GAS and they took antibiotics, or if their throat swab was negative for GAS and they did NOT take antibiotics, antibiotic treatment will be deemed 'appropriate.' All other scenarios will be deemed not 'appropriate.'

SECONDARY OUTCOMES:
Time to resolution of symptoms | 3-5 and 7-10 days post-enrolment
Caregiver satisfaction with testing | 3-5 days post-enrolment
  Likert scale
Number of days of missed school/daycare | 3-5 and 7-10 days post-enrolment
Number of days of missed work (caregiver) | 3-5 and 7-10 days post-enrolment
Number of healthcare visits for pharyngitis or sinopulmonary infections | 7 days post-enrolment
ED MD satisfaction with testing | At enrolment
  The MD who clinically assessed the patient and who later discharged the patient home will be asked - if the participant was randomized to rapid testing - whether the testing was helpful. (The outcome will be ordinal on a Likert scale). If the participant was randomized to standard testing, they will be asked how helpful NOT having rapid testing was, again measured on the same Likert scale.
Number of household contacts subsequently diagnosed with GAS pharyngitis | 7-10 days post-enrolment
Proportion of point-of-care GAS tests that are uninterpretable | at enrolment
Time required to utilize point-of-care testing | at enrolment
  Time from consent to discharge from the ED

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pernica JM, Smaill F, Kam AJ, Bartholomew A, Doan Q, Smieja M, Khan S, Sung M, Thabane L, Goldfarb DM. Single-centre, open-label, randomised, trial to compare rapid molecular point-of-care streptococcal testing to standard laboratory-based testing for the management of streptococcal pharyngitis in children: study protocol. BMJ Open. 2021 Aug 11;11(8):e047271. doi: 10.1136/bmjopen-2020-047271. PMID 34380724